CLINICAL TRIAL: NCT06563830
Title: Evaluation of the Training Applied to Nurses Prevent Medical Device-Related Pressure Injury
Brief Title: Prevent Medical Device-Related Pressure Injury
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tepecik Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Zilan BARAN, Nurse, Tepecik Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Dokuz Eylul University NURSING
Record Dates: First submitted 2024-08-08; First posted 2024-08-21 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Medical Device Site Injury; Pressure Injury
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Intervention Model Description: It is planned to conduct the study as a semi-experimental, single-group pre-test-post-test.
Masking Description: The three months incidence of medical device-related pressure injuries of patients admitted to intensive care before and after the training will be examined. At this stage, it will be conducted by two independent observers. Simultaneous monitoring will be carried out during the first week, and the harmony between the observers will be evaluated by a third party, and it will be ensured that the observations are measured Decently with the same standard. However, the bias will be reduced by having different people enter the data of the research and analyze the data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evaluation of MRRPI knowledge and attitude levels of nurses (Other): Before the training application, the effectiveness of the training application will be evaluated by applying pre-test and training application followed by two patients and intermittent post-test after three months.
  Interventions: Other: educational application

INTERVENTIONS:
Other: educational application — The content of the training to be applied to nurses will include: definition of MDRPI, etiology, prevalence and cost, staging, risk factors, nursing initiatives to be implemented to prevent MDRPI.

SUMMARY:
Medical Device-Related Pressure Injury (MDRPI) is a localized skin and/or subcutaneous tissue injury that occurs due to the pressure exerted by devices used for diagnostic or therapeutic purposes, taking the form of the medical device used. Medical device-related pressure injuries are an important adverse event with a high incidence and prevalence both in our country and in the world, accounting for more than 30% of hospital-related injuries. Medical device-related pressure injury significantly affects the quality of life of patients, but also negatively affects the cost of care for both the patient and providers. Although the most important task in preventing medical device-related pressure injuries falls on nurses, it is quite noticeable that nurses' knowledge levels of MDRPI are low in the studies conducted. MDRPI is an important issue that is ignored in nursing education and work areas in our country. In order to prevent pressure injuries associated with medical devices, it is necessary to invest more in early detection of MDRPI and improving the quality of care, studies including MDRPI risk assessment and reporting strategies are needed. In the project to be carried out in this context, it is aimed to evaluate the impact of training applied to nurses to prevent MDRPI.

DETAILED DESCRIPTION:
Medical Device-Related Pressure Injury account for more than 30% of hospital-related injuries and their incidence has been increasing steadily in recent years. According to the meta-analysis studies (n:126.150 ) the pooled incidence of MDRPI was found to be 12% (95% Cl 8-18) and the pooled prevalence of MDRPIwas found to be 10% (95% Cl 6-16). As can be seen, MDRPI is an important adverse event with a high incidence and prevalence in the world. Despite this, it is known that the MDRPI risk assessment and reporting system is used only in developed countries such as the United Kingdom, the USA and Canada on a limited basis. Medical device-related pressure injury significantly affects the quality of life of patients, but also negatively affects the cost of care for both the patient and providers. Although the incidence rate of MDRPI is high, the fact that nurses have a low level of MDRPI knowledge draws attention to the importance that should be shown to this issue. In the studies conducted, it is emphasized that in order to prevent MDRPI, more investments should be made in early detection of MDRPI and improvement of the quality of care, and studies including MDRPI risk assessment and reporting strategies are needed.

MDRPI is an important issue that is ignored in nursing education and work areas. The most important task in preventing The most important task in preventing TCIBI falls on nurses. Because patients who are at risk for the development of MDRPI need to be closely monitored continuously and prevention initiatives are needed. In this context, it is extremely important for nurses to have knowledge about the subject and to have up-to-date and evidence-based information in order to prevent MDRPI. However, when the literature is examined, it is seen that the studies measuring nurses' MDRPI knowledge are limited. In the studies conducted, it was found that nurses' knowledge levels about MDRPI were low falls on nurses. Because patients who are at risk for the development of MDRPI need to be closely monitored continuously and prevention initiatives are needed. In this context, it is extremely important for nurses to have knowledge about the subject and to have up-to-date and evidence-based information in order to prevent MDRPI. However, when the literature is examined, it is seen that the studies measuring nurses' MDRPI knowledge are limited. In the studies conducted, it was found that nurses' knowledge levels about MDRPI were low. Although its prevalence is high, education, risk assessment, reporting, prevention strategies about MDRPI are very inadequate and evidence-based studies are needed.

In this study, it was aimed to evaluate the effect of training applied to nurses to prevent MDRPI The hypotheses of the study:

H1: The MDRPI knowledge level of nurses is low before the training application.

H2: The incidence of MDRPI is high before the training application.

H03: There is no Deciency between the knowledge levels of nurses before and after the training application.

H4: Training application increases the knowledge level of nurses about MDRPI.

H5: Training application reduces the incidence of MDRPI.

H6: As the level of knowledge of MDRPI of nurses increases, the incidence of MDRPI also increases.

ELIGIBILITY:
Although the web-based training to be given within the scope of the study is applied to nurses, the results will be evaluated on both nurses and patient care results. For this reason, both nurses and intensive care inpatients constitute the sample group.

Inclusion Criteria:

Criteria for inclusion of nurses:

-Volunteer

Criteria for inclusion of patients:

* Volunteer
* Who has been hospitalized in intensive care for at least 24 hours
* Do not have a pressure injury during admission to intensive care

Exclusion Criteria:

Exclusion criteria for nurses:

-Do not volunteer

Criteria for inclusion of patients:

* Do not volunteer
* Was admitted to intensive care in less than 24 hours and transferred
* Patients with pressure injuries during admission to intensive care

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
The Incidence of Medical Device-Related Pressure Injury | Three months before the training was conducted
  The incidence of patients hospitalized in intensive care will be determined first in the study. For this purpose, patients will be observed at the same time every day during their stay in intensive care. The researcher will fill out the "MDRPI Daily Follow-up Form" for each patient who meets the inclusion criteria during hospitalization. This form has been created by the researchers in accordance with the literature information. 10 Expert opinions will be submitted before the study is carried out.
The Incidence of Medical Device-Related Pressure Injury | Three months before the training was conducted
  The incidence of patients hospitalized in intensive care will be determined first in the study. For this purpose, patients will be observed at the same time every day during their stay in intensive care. If the resulting injury develops, the "Medical Device-Related Pressure Injury Registration Form" will be used and patient monitoring will be continued for wound monitoring and other injuries. Medical Device-Related Pressure Injury Registration Form: It has been created by the researchers in accordance with the literature information. 10 Expert opinions will be submitted before the study is carried out.
Nurse's Knowledge About Medical Device-Related Pressure Injury | within three months prior to the implementation of training
  Pre-test application will be made with the "MDRPI Knowledge Scale" to determine the level of knowledge and attitude of nurses related to medical device pressure injury before training. Medical Device-related Pressure Injury Information Scale: The Confirmatory Factor Analysis (CFA) fit indices of the scale consisting of five sub-dimensions with Exploratory Factor Analysis (EFA) were determined as x2= 1.84; RMSEA= 0.05; CFI= 0.91; GFI= 0.92; AGFI= 0.90; RFI= 0.89. In addition, the total Cronbach alpha coefficient of the scale was found to be 0.798 and the test-retest score was 0.94. The lowest score that can be taken from the scale is 0 and the highest score is 25. The increase in the score indicates that the level of knowledge of TCIBY of nurses has increased.
Nurse's Attitude About Medical Device-Related Pressure Injury | within three months prior to the implementation of training
  Pre-test application will be made with "The Attidute Towards Medical Device Related Pressure Injuries" to determine the level of attitude of nurses related to medical device pressure injury before training. Preventing Medical Device-Related Pressure Injury: The Scope Validity Index of the questionnaire was found to be 98.03%, the Cronbach α value was 0.92 and the test-retest score was 0.874. The lowest score that can be obtained is 11, the highest score is 55, and the high score indicates a positive attitude towards the care and prevention of pressure injuries associated with a medical vehicle. 11 to 25 points, indicates a negative attitude towards the care and prevention of medical vehicle-related pressure injuries, a neutral attitude of 26 to 40 points, and a positive attitude of 41 to 55 points.

SECONDARY OUTCOMES:
Decrease in the Incidence of Medical Device-Related Pressure Injury | The first three months after the training application
  In order to determine the effectiveness of the training applied to nurses, the MDRPI incidence of the patients will be determined after the training and compared with the first trimester incidence. For this purpose, patients will be observed at the same time every day during their stay in intensive care. If the resulting injury develops, the "Medical Device-Related Pressure Injury Registration Form" will be used and patient monitoring will be continued for wound monitoring and other injuries.
  Medical Device-Related Pressure Injury Registration Form: It has been created by the researchers in accordance with the literature information. 10 Expert opinions will be submitted before the study is carried out.
Decrease in the Incidence of Medical Device-Related Pressure Injury | The first three months after the training application
  In order to determine the effectiveness of the training applied to nurses, the MDRPI incidence of the patients will be determined after the training and compared with the first trimester incidence. For this purpose, patients will be observed at the same time every day during their stay in intensive care. The researcher will fill out the "Medical Device-Related Pressure Injury Daily Follow-up Form" for each patient who meets the inclusion criteria during hospitalization.
  Medical Device-Related Pressure Injury Follow-up Form It has been created by the researchers in accordance with the literature information. 10 Expert opinions will be submitted before the study is carried out.

OTHER OUTCOMES:
Nurse's Knowledge About Medical Device-Related Pressure Injury | In the second and thirteenth weeks after the training
  In the second and thirteenth weeks after the training, nurses will be applied with the "MDRPI Knowledge Scale" to determine the level of knowledge of medical device-related pressure injury. Medical Device-related Pressure Injury Information Scale: The Confirmatory Factor Analysis (CFA) fit indices of the scale consisting of five sub-dimensions with Exploratory Factor Analysis (EFA) were determined as x2= 1.84; RMSEA= 0.05; CFI= 0.91; GFI= 0.92; AGFI= 0.90; RFI= 0.89. In addition, the total Cronbach alpha coefficient of the scale was found to be 0.798 and the test-retest score was 0.94. The lowest score that can be taken from the scale is 0 and the highest score is 25. The increase in the score indicates that the level of knowledge of TCIBY of nurses has increased.
Nurse's Attitude About Medical Device-Related Pressure Injury | In the second and thirteenth weeks after the training
  In the second and thirteenth weeks after the training, nurses will be applied with "The Attidute Towards Medical Device Related Pressure Injuries" to determine the level of knowledge and attitude of medical device-related pressure injury. The Attitude Scale for Preventing Medical Device-Related Pressure Injury: The Scope Validity Index of the questionnaire was found to be 98.03%, the Cronbach α value was 0.92 and the test-retest score was 0.874. The lowest score that can be obtained is 11, the highest score is 55, and the high score indicates a positive attitude towards the care and prevention of pressure injuries associated with a medical vehicle. 11 to 25 points, indicates a negative attitude towards the care and prevention of medical vehicle-related pressure injuries, a neutral attitude of 26 to 40 points, and a positive attitude of 41 to 55 points.

REFERENCES:
- [Background] Kucukkelepce GE, Karaca T, Ozkan SA. The attitude towards Medical Device-Related Pressure Injuries Questionnaire: a Turkish validity and reliability study. Wound Manag Prev. 2023 Nov;69(4):10-17. doi: 10.25270/wmp.22099. PMID 38090951
- [Result] Baran Z, Ozden D. Retrospective investigation of pressure injury in COVID-19 patients followed on invasive mechanical ventilator support. J Tissue Viability. 2024 Feb;33(1):144-149. doi: 10.1016/j.jtv.2023.10.001. Epub 2023 Oct 11. PMID 38184472
- [Result] Baran, Z., & Özden, D. (2024). Tıbbi Cihaz İlişkili Basınç Yaralanması Bilgi Ölçeği'nin Türkçe Geçerlik ve Güvenirlik Çalışması. İzmir Katip Çelebi Üniversitesi Sağlık Bilimleri Fakültesi Dergisi, 9(1), 73-80. https://doi.org/10.61399/ikcusbfd.1356400
- See also: Related Info — https://doi.org/10.61399/ikcusbfd.1356400